CLINICAL TRIAL: NCT03892161
Title: Clinical Evaluation of Adjusted Doses of Darunavir/Ritonavir With Rifampicin in HIV-infected Volunteers
Acronym: Darifi
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Risks to participation
Sponsor: University of Cape Town (Other)
Collaborators: Wits Reproductive Health and HIV Institute (Other); Desmond Tutu HIV Centre (Other)
Responsible Party: Principal Investigator, Helen Margaret McIlleron, Professor, University of Cape Town
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: Darifi
Record Dates: First submitted 2018-04-23; First posted 2019-03-27 (Actual); Last update posted 2019-04-03 (Actual); Status verified 2019-04

CONDITIONS: HIV Infections
MeSH Terms: conditions — HIV Infections | interventions — Darunavir; Ritonavir; Tablets; Rifampin; dolutegravir

STUDY DESIGN:
Intervention Model Description: A phase I, open-label, cross-over, single center, PK drug-drug interaction study will be conducted in 24 medically stable HIV-1 infected adults with viral suppression (viral load <50 copies/mL).
Who Masked: Participant, Care Provider, Investigator
Masking Description: Eligible volunteers will be switched from their standard of care PI to DRV/r 800/100 mg daily, and intensive sampling for measurement of drug concentrations will be performed at steady state. Rifampicin (600-750 mg daily depending on body weight) will then be started and subsequently the protease inhibitor doses escalated to DRV/r 1600/200 mg daily (participants randomized to arm A), OR 800/100 mg 12-hourly (arm B) for 7 days, after which patients will be switched from the daily to the 12-hourly dosing schedule (arm A) or vice versa (arm B) for a further 7 days. Rifampicin will then be stopped but the increased doses of DRV/r will be continued for a further week, before participants are switched back to their standard-of-care ART regimen. Dolutegravir (DTG) 50 mg twice daily (the dose which overcomes any interaction with rifampicin (Dooley 2013) will be added to minimize the risk of viral rebound due to possible suboptimal protease inhibitor exposures during the study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Standard dose DRV/r (Experimental): Standard dose DRV/r 800/100mg without Rifampicin
  Interventions: Drug: Darunavir/ritonavir 800/100 mg tablet
- Standard DRV/r with Rifampicin (Experimental): Rifampicin 600mg QD will be added and darunavir/ritonavir steady state pharmacokinetic analysis will be performed.
  Interventions: Drug: Darunavir/ritonavir 800/100 mg tablet; Drug: Rifampicin 600mg QD tablet and DTG 50mg BD
- Boosed ritonavir 200mg (Experimental): Rifampicin 600mg QD continued with ritonavir 200mg dose doubled QD and darunavir remains 800mg QD. The darunavir/ritonavir steady state pharmacokinetic analysis will be performed and compared.
  Interventions: Drug: Darunavir/ritonavir 800/100 mg tablet; Drug: Rifampicin 600mg QD tablet and DTG 50mg BD
- Double dose DRV/r 1600/200mg QD (Experimental): Rifampicin 600mg QD and DTG QD continued. Double dose DRV/r QD. The darunavir/ritonavir steady state pharmacokinetic analysis will be performed and compared.
  Interventions: Drug: Darunavir/ritonavir 800/100 mg tablet; Drug: Rifampicin 600mg QD tablet and DTG 50mg BD
- Double dose DRV/r 800/100mg BD (Experimental): Rifampicin 600mg QD and DTG BD continued. Double dose DRV/r QD. The darunavir/ritonavir steady state pharmacokinetic analysis will be performed and compared.
  Interventions: Drug: Darunavir/ritonavir 800/100 mg tablet; Drug: Rifampicin 600mg QD tablet and DTG 50mg BD

INTERVENTIONS:
Drug: Darunavir/ritonavir 800/100 mg tablet — Standard dose DRV/r administered
Drug: Rifampicin 600mg QD tablet and DTG 50mg BD — Rifampicin and DTG added
  Arms: Boosed ritonavir 200mg; Double dose DRV/r 1600/200mg QD; Double dose DRV/r 800/100mg BD; Standard DRV/r with Rifampicin

SUMMARY:
The DaRifi study aims:

1. Develop adjusted doses of darunavir/ritonavir for use in HIV-infected patients requiring co-treatment of TB with a rifampicin-based regimen.
2. Compare the steady state pharmacokinetics of doubled doses of DRV/r with rifampicin (in once daily and 12-hourly approaches) to standard daily doses without rifampicin.
3. Twenty-eight volunteers will be enrolled for a target of 24 participants completing the study.

DETAILED DESCRIPTION:
A significant barrier to the use of better tolerated antiretrovirals in many low-to-middle income countries (LMIC), where tuberculosis (TB) is endemic, is a lack of evidence to support their use in patients with TB. Access to optimal protease inhibitor (PI)-based regimens for patients with and without TB is urgent. Switching rifampicin to rifabutin, a weak inducer that does not significantly reduce PI concentrations, is recommended in high income countries for patients on boosted PIs who develop TB. However, rifabutin is not available in most LMIC where TB is typically treated with fixed dose combination tablets.

We will enrol virologically suppressed participants on a second-line DRV/r regimen without TB. Based on data from a Physiologically-Based PK model, we selected two adjusted doses of DRV/r (1600/200 mg daily and 800/100 mg 12 hourly) with RIF for comparison to plasma exposures with DRV/r 800/100 mg daily without RIF, in a cross-over design.

Baseline DRV steady state PK will be determined and RIF added for 7 days, then the dose of ritonavir will be increased to 200 mg; 7 days later the dose of DRV will be increased; after another 7 days participants will be crossed over to the alternative adjusted DRV dose.

DRV will be measured in plasma samples after observed doses at baseline and after each dose adjustment. Non-compartmental analysis will be used to estimate the PK measures. Clinical adverse events, ALT, and bilirubin will be monitored every 2 to 3 days during treatment with RIF.

ELIGIBILITY:
Inclusion Criteria

* Male or female
* Aged 18 to 60 years, inclusive
* Weighing > 38 kg
* BMI > 18.5 kg/m2
* HIV-1 infected
* HIV-1 RNA <50 copies/mL
* CD4+ lymphocyte count > 200 cells/L
* C-reactive protein <10 mg/L
* Established on current ART regimen of boosted protease inhibitor plus 2 NRTIs for at least 3 months.
* Women must be postmenopausal, surgically sterile or practicing an effective birth control method (established before and maintained throughout the trial). Women who are not sexually active must agree to use an effective birth control method if they become heterosexually active during the trial.
* Understand the purpose of and procedures required for the study and having confirmed they are willing to participate in the study by signing the informed consent document.

Exclusion criteria (volunteers meeting any of the criteria will be excluded)

* TB (confirmed or suspected)
* Any symptoms of TB - as assessed by the WHO symptom-screening algorithm: self-reported or documented weight loss, cough, night sweats or fever.
* Clinical or laboratory evidence of significantly impaired hepatic function, or documented hepatic cirrhosis
* Clinical or laboratory evidence of acute viral hepatitis
* Co-infected with HBV or HCV.
* ALT grade 2 or higher (as defined by DAIDS grading table (ALT >2.5 x ULN)
* DAIDS grade 3 or 4 laboratory abnormality
* Active (not clinically stabilized >4 weeks) AIDS defining illness (Category C conditions according to the Center for Disease Control Classification System for HIV infection) with the following exceptions:
* Stable cutaneous Kaposi's Sarcoma (no internal organ involvement other than oral lesions) that is unlikely to require any form of systemic therapy during the study.
* Estimated creatinine clearance <50 mL/min.
* Active clinically significant renal or gastro-intestinal disease.
* Any active clinically significant or life-threatening disease, medical or psychiatric condition, or findings during screening, that in the investigator's opinion would compromise the safety of the participant or the study outcome, or their ability to comply with the study procedures.
* Chronic medical requirement for any drugs that are known to affect the PK of the study drugs.
* Active drug/alcohol abuser.
* Pregnant or breastfeeding.
* Increased risks of drug side effects/hypersensitivity reactions e.g. haemophilia or history of sulfonamide allergy.
* Currently enrolled in an investigational drug study or has participated in an investigational drug study within the 4 weeks before screening.
* Unable to comply with peri-study restrictions

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 17 (Actual)
Dates: Start 2018-04-12 (Actual); Primary Completion 2018-11-22 (Actual); Study Completion 2018-11-22 (Actual)

PRIMARY OUTCOMES:
Darunavir plasma concentrations nanogram per milliliter (ng/ml) | 1 year
  Darunavir plasma concentrations will be compared with rifampicin and without rifampicin.

SECONDARY OUTCOMES:
Alanine Transaminase (ALT) blood level (iu/L) | 1 Year
  Clinical safety will be monitored, ALT liver enzyme tests will be evaluated every 3 days.

CONTACTS AND LOCATIONS:
Overall Officials: Helen McIlleron, PhD, Principal Investigator — University of Cape Town
Locations (1):
- Clinical Research Centre, Cape Town, Western Cape, South Africa

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Baietto L, Calcagno A, Motta I, Baruffi K, Poretti V, Di Perri G, Bonora S, D'Avolio A. A UPLC-MS-MS method for the simultaneous quantification of first-line antituberculars in plasma and in PBMCs. J Antimicrob Chemother. 2015 Sep;70(9):2572-5. doi: 10.1093/jac/dkv148. Epub 2015 Jun 11. PMID 26066583
- [Background] Chirehwa MT, Rustomjee R, Mthiyane T, Onyebujoh P, Smith P, McIlleron H, Denti P. Model-Based Evaluation of Higher Doses of Rifampin Using a Semimechanistic Model Incorporating Autoinduction and Saturation of Hepatic Extraction. Antimicrob Agents Chemother. 2015 Nov 9;60(1):487-94. doi: 10.1128/AAC.01830-15. Print 2016 Jan. PMID 26552972
- [Background] D'Avolio A, Simiele M, Siccardi M, Baietto L, Sciandra M, Oddone V, Stefani FR, Agati S, Cusato J, Bonora S, Di Perri G. A HPLC-MS method for the simultaneous quantification of fourteen antiretroviral agents in peripheral blood mononuclear cell of HIV infected patients optimized using medium corpuscular volume evaluation. J Pharm Biomed Anal. 2011 Mar 25;54(4):779-88. doi: 10.1016/j.jpba.2010.10.011. Epub 2010 Nov 10. PMID 21071165
- [Background] Decloedt EH, McIlleron H, Smith P, Merry C, Orrell C, Maartens G. Pharmacokinetics of lopinavir in HIV-infected adults receiving rifampin with adjusted doses of lopinavir-ritonavir tablets. Antimicrob Agents Chemother. 2011 Jul;55(7):3195-200. doi: 10.1128/AAC.01598-10. Epub 2011 May 2. PMID 21537021
- [Background] Decloedt EH, Maartens G, Smith P, Merry C, Bango F, McIlleron H. The safety, effectiveness and concentrations of adjusted lopinavir/ritonavir in HIV-infected adults on rifampicin-based antitubercular therapy. PLoS One. 2012;7(3):e32173. doi: 10.1371/journal.pone.0032173. Epub 2012 Mar 7. PMID 22412856
- [Background] De Nicolo A, Bonifacio G, Boglione L, Cusato J, Pensi D, Tomasello C, Di Perri G, D'Avolio A. UHPLC-MS/MS method with automated on-line solid phase extraction for the quantification of entecavir in peripheral blood mononuclear cells of HBV+ patients. J Pharm Biomed Anal. 2016 Jan 25;118:64-69. doi: 10.1016/j.jpba.2015.10.017. Epub 2015 Oct 22. PMID 26517850
- [Background] Dooley KE, Sayre P, Borland J, Purdy E, Chen S, Song I, Peppercorn A, Everts S, Piscitelli S, Flexner C. Safety, tolerability, and pharmacokinetics of the HIV integrase inhibitor dolutegravir given twice daily with rifampin or once daily with rifabutin: results of a phase 1 study among healthy subjects. J Acquir Immune Defic Syndr. 2013 Jan 1;62(1):21-7. doi: 10.1097/QAI.0b013e318276cda9. PMID 23075918
- [Background] Haas DW, Koletar SL, Laughlin L, Kendall MA, Suckow C, Gerber JG, Zolopa AR, Bertz R, Child MJ, Hosey L, Alston-Smith B, Acosta EP; A5213 StudyTeam. Hepatotoxicity and gastrointestinal intolerance when healthy volunteers taking rifampin add twice-daily atazanavir and ritonavir. J Acquir Immune Defic Syndr. 2009 Mar 1;50(3):290-3. doi: 10.1097/QAI.0b013e318189a7df. PMID 19194314
- [Background] la Porte CJ, Colbers EP, Bertz R, Voncken DS, Wikstrom K, Boeree MJ, Koopmans PP, Hekster YA, Burger DM. Pharmacokinetics of adjusted-dose lopinavir-ritonavir combined with rifampin in healthy volunteers. Antimicrob Agents Chemother. 2004 May;48(5):1553-60. doi: 10.1128/AAC.48.5.1553-1560.2004. PMID 15105105
- [Background] L'homme RF, Nijland HM, Gras L, Aarnoutse RE, van Crevel R, Boeree M, Brinkman K, Prins JM, Juttmann JR, Burger DM. Clinical experience with the combined use of lopinavir/ritonavir and rifampicin. AIDS. 2009 Apr 27;23(7):863-5. doi: 10.1097/QAD.0b013e328329148e. PMID 19352137
- [Background] Nijland HM, L'homme RF, Rongen GA, van Uden P, van Crevel R, Boeree MJ, Aarnoutse RE, Koopmans PP, Burger DM. High incidence of adverse events in healthy volunteers receiving rifampicin and adjusted doses of lopinavir/ritonavir tablets. AIDS. 2008 May 11;22(8):931-5. doi: 10.1097/QAD.0b013e3282faa71e. PMID 18453852
- [Background] Panel on Antiretroviral Guidelines for Adults and Adolescents. Guidelines for the use of antiretroviral agents in HIV-1-infected adults and adolescents. Department of Health and Human Services. http://www.aidsinfo.nih.gov/ContentFiles/AdultandAdolescentGL.pdf
- [Background] Rabie et al., Pharmacokinetics of lopinavir/ritonavir superboosting in infants and young children co-infected with HIV and TB. 7th Int WS on HIV Pediatrics 2015, Vancouver
- [Background] Ren Y, Nuttall JJ, Egbers C, Eley BS, Meyers TM, Smith PJ, Maartens G, McIlleron HM. Effect of rifampicin on lopinavir pharmacokinetics in HIV-infected children with tuberculosis. J Acquir Immune Defic Syndr. 2008 Apr 15;47(5):566-9. doi: 10.1097/QAI.0b013e3181642257. PMID 18197120
- [Background] Roberts O, Khoo S, Owen A, Siccardi M. Interaction of Rifampin and Darunavir-Ritonavir or Darunavir-Cobicistat In Vitro. Antimicrob Agents Chemother. 2017 Apr 24;61(5):e01776-16. doi: 10.1128/AAC.01776-16. Print 2017 May. PMID 28193650
- [Background] Sekar VJ, Lefebvre E, De Pauw M, Vangeneugden T, Hoetelmans RM. Pharmacokinetics of darunavir/ritonavir and ketoconazole following co-administration in HIV-healthy volunteers. Br J Clin Pharmacol. 2008 Aug;66(2):215-21. doi: 10.1111/j.1365-2125.2008.03191.x. Epub 2008 Apr 8. PMID 18460033
- [Background] Sekar V, Lefebvre E, De Marez T, De Pauw M, De Paepe E, Vangeneugden T, Hoetelmans RM. Pharmacokinetic interaction between indinavir and darunavir with low-dose ritonavir in healthy volunteers. Intervirology. 2010;53(3):176-82. doi: 10.1159/000289341. Epub 2010 Mar 3. PMID 20197684
- [Background] Sekar V, Lavreys L, Van de Casteele T, Berckmans C, Spinosa-Guzman S, Vangeneugden T, De Pauw M, Hoetelmans R. Pharmacokinetics of darunavir/ritonavir and rifabutin coadministered in HIV-negative healthy volunteers. Antimicrob Agents Chemother. 2010 Oct;54(10):4440-5. doi: 10.1128/AAC.01749-09. Epub 2010 Jul 26. PMID 20660678
- [Background] Siccardi, et al. In Silico Simulation of Interaction Between Rifampicin and Boosted Darunavir. Conference on Retroviruses and opportunistic infections, abstr: 532. Seattle 2015.
- [Background] Soon GH, Shen P, Yong EL, Pham P, Flexner C, Lee L. Pharmacokinetics of darunavir at 900 milligrams and ritonavir at 100 milligrams once daily when coadministered with efavirenz at 600 milligrams once daily in healthy volunteers. Antimicrob Agents Chemother. 2010 Jul;54(7):2775-80. doi: 10.1128/AAC.01564-09. Epub 2010 Apr 12. PMID 20385850
- [Background] Sunpath H, Winternheimer P, Cohen S, Tennant I, Chelin N, Gandhi RT, Murphy RA. Double-dose lopinavir-ritonavir in combination with rifampicin-based anti-tuberculosis treatment in South Africa. Int J Tuberc Lung Dis. 2014 Jun;18(6):689-93. doi: 10.5588/ijtld.13.0492. PMID 24903940
- [Background] Zhang C, McIlleron H, Ren Y, van der Walt JS, Karlsson MO, Simonsson US, Denti P. Population pharmacokinetics of lopinavir and ritonavir in combination with rifampicin-based antitubercular treatment in HIV-infected children. Antivir Ther. 2012;17(1):25-33. doi: 10.3851/IMP1915. PMID 22267466
- [Background] Zhang C, Denti P, Decloedt EH, Ren Y, Karlsson MO, McIlleron H. Model-based evaluation of the pharmacokinetic differences between adults and children for lopinavir and ritonavir in combination with rifampicin. Br J Clin Pharmacol. 2013 Nov;76(5):741-51. doi: 10.1111/bcp.12101. PMID 23432610
- [Background] Zhang C, Denti P, Decloedt E, Maartens G, Karlsson MO, Simonsson US, McIlleron H. Model-based approach to dose optimization of lopinavir/ritonavir when co-administered with rifampicin. Br J Clin Pharmacol. 2012 May;73(5):758-67. doi: 10.1111/j.1365-2125.2011.04154.x. PMID 22126409
- [Derived] De Nicolo A, Calcagno A, Motta I, De Vivo E, D'Avolio A, Di Perri G, Wiesner L, Ebrahim IE, Maartens G, Orrell C, McIlleron H. The Effect of Rifampicin on Darunavir, Ritonavir, and Dolutegravir Exposure within Peripheral Blood Mononuclear Cells: a Dose Escalation Study. Antimicrob Agents Chemother. 2022 Jun 21;66(6):e0013622. doi: 10.1128/aac.00136-22. Epub 2022 May 18. PMID 35583344